CLINICAL TRIAL: NCT01891409
Title: Use of the Shang Ring Device in All Four Childhood Age Groups in the African Population
Brief Title: Use of the Shang Ring Circumcision Device in Boys Below 18 Years Old in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EngenderHealth (Other)
Collaborators: Weill Medical College of Cornell University (Other); Kenya National AIDS & STI Control Programme (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCC-0139-01; GCC-0139 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV prevention; Male Circumcision; Children; Childhood; Shang Ring
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Single arm study study for use of Shang Ring device for male circumcision in children
  Interventions: Device: Male circumcision using the Shang Ring device

INTERVENTIONS:
Device: Male circumcision using the Shang Ring device
  Other Names: Shang ring male circumcision device

SUMMARY:
A proof of concept study to evaluate the feasibility of using the Shang Ring, a novel male circumcision device across all childhood age groups namely infants (under 1), 1-5 age group, 6-12 age group and the 13-17 age group. The study will evaluate the safety, efficacy and course of wound healing when using the Shang Ring technique across the four childhood age groups.

DETAILED DESCRIPTION:
A proof of concept study to evaluate the feasibility of using the Shang Ring, a novel male circumcision device across all childhood age groups namely infants (under 1), 1-5 age group, 6-12 age group and the 13-17 age group. The study will evaluate efficacy, procedure time, difficulties during surgery and post-operative events shall be assessed. To evaluate safety, the investigators will clinically observe for adverse events during the course of healing. The investigators will also evaluate to length of time taken for complete healing to be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Must be accompanied by the parent or legally acceptable representative (LAR), who freely consents for participation of the child into the study;
* Assent from participant 7 years of age and above who understand study procedure;
* Aged between 1 month and 17 years(inclusive);
* Body weight of more than 2.5 kgs and penile shaft more than 1 cm in length.
* Must be in good general health;
* Must be free of genital ulcerations or other visible signs of STI (on examination);
* Parent or LAR and if possible the client must be able to understand study procedures and requirements of study participation;
* Parent or LAR must agree to return the client to the study site for the full schedule of follow-up visits after his circumcision;
* Parent or LAR must have a cell phone or access to a cell phone; and,
* Parent or LAR must agree to provide the study staff with an address, phone number, or other locator information while participating in the research study.

Exclusion Criteria:

* Has a known allergy or sensitivity to lidocaine or other local anesthesia;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
* Has known bleeding/clotting disorder (e.g. hemophilia);
* Has any congenital genitourinary abnormality;
* Has an active genital infection, anatomic abnormality or other condition (e.g. severe obesity, diabetes or sickle cell anemia), which in the opinion of the surgeon, prevents the man from undergoing a circumcision as part of this study; or
* Is currently participating in another biomedical research study.

Ages: 1 Month to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate safety when using the Shang Ring technique across the 4 age groups ranging from infants to adolescents. | 42 days after circumcision
  Documentation of adverse events based on clinical exam findings

SECONDARY OUTCOMES:
To evaluate efficacy when using the Shang Ring technique across the 4 age groups ranging from infants to adolescents. | 42 days after circumcision
  To evaluate efficacy, procedure time, peri- and postoperative surgical complications, and problems with use of the device will be assessed.
To evaluate the course of wound healing when using the Shang Ring technique across the 4 age groups ranging from infants to adolescents. | 42 days after circumcision
  Evaluation of the course of healing and length of time required for complete healing will be based on clinical exam findings.
To determine the acceptability of the Shang Ring device by the participants (or their parents) | 42 days after circumcison
  Clients and/or parents shall be interviewed on their experience with the Shang Ring during their participation in the study.
To evaluate the ease of use of the Shang Ring technique across the 4 age groups ranging from infants to adolescents | 42 days after circumcision
  To evaluate the ease of use of the Shang Ring device, clinicians shall be interviewed on the difficulties they faced with using the device and their perception about use of the device relative to conventional surgical approaches

CONTACTS AND LOCATIONS:
Overall Officials: Quentin Awori, MBChB, CPI, Principal Investigator — EngenderHealth
Locations (1):
- Homa Bay District Hospital, Homa Bay, Kenya